CLINICAL TRIAL: NCT01928576
Title: A Phase II Study of Epigenetic Therapy With Azacitidine and Entinostat With Concurrent Nivolumab in Subjects With Metastatic Non-Small Cell Lung Cancer.
Brief Title: Phase II Anti-PD1 Epigenetic Therapy Study in NSCLC.
Acronym: NA_00084192
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Rising Tide Foundation (Other); Stand Up To Cancer (Other); Bristol-Myers Squibb (Industry); Celgene (Industry); Syndax Pharmaceuticals (Industry); Rhone-Poulenc Rorer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1353; NA_00084192 (Other: JHMIRB); 119134 (Other Grant/Funding Number: Rising Tide Foundation); 117207 (Other Grant/Funding Number: Stand Up To Cancer); 121445 (Other Grant/Funding Number: JH FAMRI); 119134 (Other Grant/Funding Number: Rhone-Poulenc ROrer); CA209-117 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer; Epigenetic Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Azacitidine; entinostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm C (Experimental): Nivolumab 3mg/kg every 2 weeks until progression
  Interventions: Drug: Nivolumab
- Arm D (Experimental): Anti-PD-1/PD-L1 treatment naïve patients only
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Drug: Nivolumab
- Arm E (Experimental): Patients must have had refractory (Arm E=less than 24 weeks from first dose of anti-PD-1/PD-L1) disease during or after anti-PD-1 or anti-PD-L1 therapy and, in the opinion of the investigator, must be unlikely to benefit from nivolumab monotherapy.
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Drug: Nivolumab
- Arm F (Experimental): Patients must have had recurrent (Arm F=more than 24 weeks from first dose of anti-PD1/PD-L1) disease during or after anti-PD-1 or anti-PD-L1 therapy and, in the opinion of the investigator, must be unlikely to benefit from nivolumab monotherapy.
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Interventions: Drug: Azacitidine; Drug: Entinostat; Drug: Nivolumab
- Arm A (Experimental): Anti-PD-1/PD-L1 treatment naïve patients only Every 28 days for 2 cycles Azacitidine 40mg/m2 subcutaneous days 1-6 and 8-10 Entinostat 7mg by mouth Days 3 and 10
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg
  Interventions: Drug: Azacitidine; Drug: Entinostat; Drug: Nivolumab
- Arm B (Experimental): Every 28 days for 2 cycles CC-486 300 mg by mouth days 1 - 21
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Interventions: Drug: Nivolumab; Drug: CC-486 300

INTERVENTIONS:
Drug: Azacitidine
  Other Names: 5-AZA, Vidaza
  Arms: Arm A; Arm D; Arm E; Arm F
Drug: Entinostat
  Arms: Arm A; Arm D; Arm E; Arm F
Drug: Nivolumab
  Other Names: Opdivo
Drug: CC-486 300
  Arms: Arm B

SUMMARY:
Response Rate

DETAILED DESCRIPTION:
Objective response rate to Nivolumab preceded by epigenetic priming. Response will be assessed by RECIST 1.1 criteria, baseline scans for this assessment will be the baseline scans done within 4 weeks of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven stage IIIB, IV or recurrent non-small cell lung cancer. Patients must be willing to undergo a pre-treatment biopsy, either core needle biopsy or equivalent amount or via excisional specimen. (cytology specimen not acceptable for this purpose).
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease. A CT scan of the abdomen and pelvis is not required for patients with no disease in these areas.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of azacitidine with entinostat, or of Nivolumab, in patients <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Life expectancy of greater than 12 weeks.
* Patients must have adequate organ and marrow function.
* The effects of entinostat, azacitidine, and Nivolumab, on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for up to 23 weeks after the last dose of nivolumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men who are sexually active with women of childbearing potential must also use an adequate contraceptive method for up to 31 weeks after fhe last dose of nivolumab.
* Ability to understand and the willingness to sign a written informed consent document.
* All adenocarcinoma patients must be tested for ALK rearrangements and EGFR (Exon 19 Deletion and Exon 21 L8585R Substitution) mutations and must have been treated with EGFR or ALK TKI therapy if found to have an actionable alteration. If patients are KRAS positive, testing for ALK rearrangements and EGFR mutations is not applicable.
* All patients should have been offered a platinum-based chemotherapy. For EGFR/ALK wild type patients, no more than two prior chemotherapy-based lines of therapy for advanced or metastatic NSCLC is permitted. For EGFR mutated or ALK translocated patients, no more than three prior lines of therapy for advanced or metastatic NSCLC is permitted. Patients who refuse platinum based chemotherapy, may be allowed to enroll if they meet all other criteria.

  * Patients who received adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) and developed recurrent or metastatic disease within 6 months of completing therapy are eligible and the adjuvant or neoadjuvant chemotherapy will count as a line of therapy as above.
  * Subjects with recurrent disease > 6 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum-doublet regimen given to treat the recurrences, are eligible and do not count as another line of therapy for advanced disease.
  * Subjects who received pemetrexed, bevacizumab, or erlotinib as maintenance therapy (nonprogressors with platinum-based doublet chemotherapy) and subsequently progressed after maintenance therapy, are eligible and do not count as a line of therapy. However, subject who received a tyrosine kinase inhibitor after failure of a prior platinum-based therapy, that tyrosine kinase inhibitor therapy would count as an additional line of therapy.
  * Patients who have been treated with prior standard of care PD-1/L1 agents, alone or in combination with chemotherapy, are eligible. Patients previously treated on clinical trials with non PD-1/PD-L1 immunotherapy agents are eligible. Patients who have been treated with a PD-1/L1 agent in more than 1 line of therapy (as standard of care or in clinical trial) are not eligible.
* Arm-specific eligibility criteria

  * Arm D: Anti-PD-1/PD-L1 treatment naïve patients only
  * Arm E & F: Anti-PD-1/PD-L1 treatment experienced patients: Patients must have had refractory (Arm E=less than 24 weeks from first dose of anti-PD-1/PD-L1) or recurrent (Arm F=more than 24 weeks from first dose of anti-PD-1/PD-L1) disease during or after anti-PD-1 or anti-PD-L1 therapy and, in the opinion of the investigator, must be unlikely to benefit from nivolumab monotherapy.
* Patients must have disease amenable to biopsy at the time of enrollment as biopsies are required for study participation.

Exclusion Criteria:

* Any active history of a known autoimmune disease. Subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a history of interstitial lung disease that has required intubation in the past (i.e. such as Asthma or COPD).
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Patients who are receiving any other anticancer therapy.
* Patients with uncontrolled brain metastases. Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks without the use of steroids or on stable or decreasing dose of < 10mg daily prednisone (or equivalent), and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with a history of carcinomatous meningitis are not eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to entinostat, azacitidine, or Nivolumab.
* Known or suspected hypersensitivity to azacitidine or mannitol
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because entinostat, azacitidine, and Nivolumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with entinostat, azacitidine, or Nivolumab breastfeeding should be discontinued if the mother is treated on this protocol.
* HIV-positive patients are excluded. (Patients cannot have known history of HIV. Testing for it at baseline is not required unless it is suspected they may have it).
* Patients with active hepatitis B or hepatitis C are excluded. (Patients cannot have known history of hepatitis B or hepatitis C. Testing for it at baseline is not required unless it is suspected they may have it).
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Patients with malabsorption in the small intestine or other conditions that would preclude administration of oral medication.
* Prior therapy with DNA methyltransferase therapy or HDAC inhibitor therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Julie Brahmer, MD, Baltimore, Maryland
  - UPMC Cancer Center- Hillman Cancer Center, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 patients were not eligible. The list of reasons for subjects not being eligible include Subject had did not have disease amenable to biopsy, Disease Progression, elevated creatinine, COVID-19, hyponatremia, patient declined, patient sent to hospice, deceased, history of pneumonitis, not have enough tissue for biopsy, central nervous system involvement, pericardial effusion, brain metastasis, and Hypoxemia.
Groups:
- Arm C: Nivolumab 3mg/kg every 2 weeks until progression
  Nivolumab
- Arm D: Anti-PD-1/PD-L1 treatment naïve patients only
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Azacitidine
  Entinostat
  Nivolumab
- Arm E: Patients must have had refractory (Arm E=less than 24 weeks from first dose of anti-PD-1/PD-L1) disease during or after anti-PD-1 or anti-PD-L1 therapy and, in the opinion of the investigator, must be unlikely to benefit from nivolumab monotherapy.
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Azacitidine
  Entinostat
  Nivolumab
- Arm F: Patients must have had recurrent (Arm F=more than 24 weeks from first dose of anti-PD1/PD-L1) disease during or after anti-PD-1 or anti-PD-L1 therapy and, in the opinion of the investigator, must be unlikely to benefit from nivolumab monotherapy.
  Every 28 days for 6 cycles Azacitidine 40mg/m2 days 1-5 and 8-10 Entinostat 5mg Days 3 and 10 Nivolumab 3mg/kg Days 1 and 15
  Followed by:
  Nivolumab 3mg/kg every 2 weeks until progression
  After a patient has completed 6 months of nivolumab, they can receive nivolumab every 4 weeks instead of every 2 weeks. The dose for Nivolumab every 4 weeks is 480mg.
  Azacitidine
  Entinostat
  Nivolumab
Period: Overall Study
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Started | 32 | 7 | 21 | 14 | 7 | 19
Completed | 32 | 7 | 21 | 14 | 7 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F | Total
Number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 19 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: age data was missing for 1 participant in Arm F.
  years
    number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 18 | 99
    (all) | 62.7 (10) | 67.3 (6.6) | 64.2 (9) | 66.7 (10.3) | 73 (9.7) | 66.6 (7.5) | 72 (9.36)
Age, Continuous [Median (Full Range); unit: years] — Population: age data was missing for 1 participant in Arm F
  years
    number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 18 | 99
    (all) | 63.5 [45 to 83] | 67 [58 to 76] | 62 [53 to 83] | 65.5 [47 to 84] | 70 [63 to 90] | 66.6 [55 to 84] | 70 [45 to 90]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Female | 16 | 4 | 9 | 5 | 3 | 8 | 45
  Male | 16 | 3 | 12 | 9 | 4 | 10 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 6 | 19 | 14 | 6 | 18 | 94
  Unknown or Not Reported | 1 | 1 | 2 | 0 | 1 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 2 | 3 | 1 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 1 | 3 | 3 | 0 | 1 | 13
  White | 21 | 4 | 14 | 9 | 6 | 15 | 69
  More than one race | 1 | 0 | 1 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 7 | 21 | 14 | 7 | 19 | 100

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Percentage of participants with response to combination Nivolumab and epigenetic therapy. Response will be assessed by RECIST 1.1 criteria, where complete response (CR)= disappearance of all target lesions, partial response (PR) is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 2 years
Population: 1 patient from ARM A and 1 patient from ARM C did not have documentation of resict reads to analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 31 | 7 | 20 | 14 | 7 | 19
Participants | 4 | 1 | 5 | 3 | 1 | 2

2. Secondary Outcome: Progression Free Survival
Description: Number of months from the time of randomization until radiologic (per RECIST 1.1) or clinical progression or death, whichever comes first.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 19
months | 4.6 [3.7 to 13.7] | 3.7 [0.9 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 5.7 [2.1 to 14.7] | 7.8 [3.2 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 4.9 [1.4 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 3.8 [2.9 to 6.64]

3. Secondary Outcome: Time to Progression
Description: Number of months from the time nivolumab begins until radiologic (per RECIST 1.1) or clinical progression is noted.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 19
months | 4.6 [3.4 to 13.7] | 3.7 [0.9 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 5.7 [2.1 to 14.7] | 7.8 [3.2 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 4.9 [1.4 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 3.8 [2.9 to 21.8]

4. Secondary Outcome: Overall Survival
Description: Number of months from the time of randomization until death. Estimation will be by the Kaplan-Meier method.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 19
months | 10.5 [7.7 to 25.1] | 4 [1.3 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 16.9 [12.9 to 57.4] | 14 [7.9 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 5 [3.2 to NA] — not estimable because the upper confidence limits for the survivor function in this cohort was never less than 50% | 12.1 [7.7 to 25.6]

5. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Dose-limiting Toxicities
Description: Number of participants who experience adverse events as defined by CTCAE v4.0 that require a dose reduction.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
Number analyzed (Participants) | 32 | 7 | 21 | 14 | 7 | 19
Participants | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All Adverse events and Serious Adverse events data was collected during the treatment phase of the study and then at a 30 day follow up visit, up to 2 years. Death assessed up to 5 years post treatment.
Arm/Group | ARM A | ARM B | Arm C | Arm D | Arm E | Arm F
All-Cause Mortality (participants affected / at risk) | 22/32 | 6/7 | 12/21 | 5/14 | 7/7 | 12/19
Serious Adverse Events (participants affected / at risk) | 4/32 | 1/7 | 1/21 | 0/14 | 2/7 | 0/19
Other Adverse Events (participants affected / at risk) | 32/32 | 7/7 | 21/21 | 14/14 | 7/7 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (N=32) | ARM B (N=7) | Arm C (N=21) | Arm D (N=14) | Arm E (N=7) | Arm F (N=19)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin T increased (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A (N=32) | ARM B (N=7) | Arm C (N=21) | Arm D (N=14) | Arm E (N=7) | Arm F (N=19)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 0 (0) | 4 (5) | 3 (7) | 0 (0) | 2 (2)
Absolute Lymphocytes Decreased (Investigations) | 3 (6) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 2 (6)
Absolute neutrophil Count (ANC)decreased (Investigations) | 2 (3) | 2 (3) | 2 (4) | 1 (1) | 0 (0) | 1 (4)
Alanine Aminotransferase Increased (Investigations) | 3 (6) | 1 (1) | 5 (14) | 2 (14) | 0 (0) | 0 (0)
albumin decreased (Investigations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
alkaline phosphae increased (Investigations) | 10 (12) | 2 (2) | 4 (4) | 9 (41) | 6 (18) | 1 (1)
Alopecia (General disorders) | 5 (5) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 0 (0)
Anemia (Investigations) | 17 (31) | 4 (9) | 10 (22) | 7 (29) | 2 (6) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 19 (34) | 5 (8) | 8 (12) | 2 (5) | 3 (4) | 5 (8)
Anxiety (Psychiatric disorders) | 4 (9) | 1 (3) | 7 (10) | 3 (5) | 0 (0) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (1) | 4 (7) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 6 (9) | 2 (3) | 3 (8) | 2 (9) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (14) | 3 (4) | 4 (4) | 1 (1) | 0 (0) | 4 (6)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (2)
Chest Pain (Non-Cardiac) (Musculoskeletal and connective tissue disorders) | 5 (9) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (4)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (30) | 5 (14) | 7 (12) | 11 (14) | 3 (4) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (27) | 4 (8) | 16 (32) | 3 (14) | 3 (6) | 6 (10)
creatine increased (Investigations) | 2 (2) | 1 (1) | 2 (5) | 1 (2) | 0 (0) | 1 (3)
Dehydration (General disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (8) | 1 (1) | 1 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 1 (2) | 9 (13) | 1 (1) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 7 (10) | 1 (4) | 3 (4) | 4 (4) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 5 (7) | 0 (0) | 3 (4) | 3 (5) | 1 (1) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
Dysguesia (Gastrointestinal disorders) | 7 (11) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Dyspepsia (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 3 (4) | 4 (5) | 2 (3) | 2 (3) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 9 (13) | 1 (1) | 3 (4) | 2 (6) | 3 (3) | 1 (2)
Fatigue (General disorders) | 26 (54) | 7 (16) | 15 (33) | 9 (16) | 5 (6) | 8 (18)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 6 (8) | 0 (0) | 3 (3) | 7 (15) | 1 (1) | 4 (7)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (11) | 0 (0) | 12 (83) | 6 (13) | 0 (0) | 2 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (9) | 0 (0) | 3 (21) | 2 (4) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (17) | 1 (3) | 7 (65) | 6 (19) | 0 (0) | 2 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (35) | 5 (9) | 10 (14) | 5 (15) | 4 (4) | 3 (7)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2) | 5 (24) | 5 (13) | 0 (0) | 0 (0)
fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 26 (54) | 7 (16) | 16 (33) | 9 (16) | 5 (6) | 8 (18)
Fever (General disorders) | 1 (2) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoalbumenia (Metabolism and nutrition disorders) | 19 (58) | 2 (5) | 15 (183) | 7 (46) | 1 (1) | 2 (13)
hypocalcemia (Metabolism and nutrition disorders) | 7 (10) | 0 (0) | 6 (18) | 4 (10) | 2 (3) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 2 (2) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (8) | 1 (1) | 6 (14) | 0 (0) | 1 (1) | 1 (3)
Hyponatrema (Metabolism and nutrition disorders) | 6 (7) | 1 (1) | 6 (9) | 4 (7) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (8) | 2 (4) | 3 (5) | 4 (12) | 0 (0) | 2 (8)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Injection site reaction (Infections and infestations) | 23 (33) | 0 (0) | 1 (2) | 4 (6) | 1 (1) | 4 (16)
Insomnia (Psychiatric disorders) | 9 (12) | 0 (0) | 3 (9) | 1 (2) | 2 (2) | 2 (2)
Oral Mucositis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (6) | 1 (1) | 1 (1) | 2 (2)
Nasuea (Gastrointestinal disorders) | 17 (28) | 4 (8) | 7 (8) | 8 (12) | 3 (5) | 8 (24)
Neutrophil count decreased (Investigations) | 6 (7) | 2 (3) | 2 (3) | 2 (3) | 0 (0) | 1 (4)
Pain (General disorders) | 8 (17) | 2 (3) | 8 (24) | 6 (11) | 5 (8) | 3 (9)
neuropathy (Nervous system disorders) | 2 (3) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 4 (4) | 1 (4) | 2 (5) | 5 (8) | 3 (4) | 1 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (17) | 0 (0) | 5 (27) | 3 (6) | 1 (1) | 7 (9)
Sore throat (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Voice Hoarseness (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 7 (11) | 2 (2) | 2 (2) | 3 (5) | 2 (3) | 4 (7)
Weight loss (Investigations) | 9 (14) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 1 (1)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 1 (3)
White Blood Cell Decreased (Investigations) | 16 (34) | 4 (19) | 7 (14) | 7 (15) | 2 (2) | 2 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT01928576/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT01928576/ICF_001.pdf